CLINICAL TRIAL: NCT00924651
Title: A Study of the Effects of Exercise on Cancer-Related Fatigue
Brief Title: Exercise in Lessening Fatigue Caused by Cancer in Patients Undergoing Chemotherapy
Acronym: EXCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Professor, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UCCO08106; URCC0701; U10CA037420 (NIH); UCCO-08106 (Other: URCC); URCC 0701 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Results first posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: fatigue; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Fatigue | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care + EXCAP (Experimental): Personalized exercise prescription
  Interventions: Behavioral: exercise
- Standard Care (No Intervention): Wait list control

INTERVENTIONS:
Behavioral: exercise — home based walking and progressive resistance training exercise
  Other Names: EXCAP
  Arms: Standard Care + EXCAP

SUMMARY:
RATIONALE: Physical activity may help lessen fatigue caused by cancer in patients receiving chemotherapy. It is not yet known whether a home-based walking and resistance-band exercise program is effective in lessening fatigue.

PURPOSE: This randomized phase III trial is studying how well exercise works in lessening fatigue caused by cancer in patients undergoing chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of a home-based walking and progressive-resistance exercise program in reducing cancer-related fatigue (CRF) in patients undergoing chemotherapy.

OUTLINE: This is a multicenter study. Patients are stratified according to participating site, chemotherapy course length (2 weeks vs 3 weeks), gender, and degree of fatigue reported on the study assessment questionnaire (≤ 5 vs > 5). Patients are randomized to 1 of 2 intervention arms.

* Arm I: Patients receive standard chemotherapy.
* Arm II: Patients receive a home-based walking kit comprising an Exercise for Cancer Patients Manual, a pedometer, and therapeutic resistance bands. Patients undergo moderately intense aerobic exercise (walking) monitored by a pedometer, and low to moderately intense progressive-resistance exercise using therapeutic resistance bands for 6 weeks. Patients also receive standard chemotherapy.

Patients in both arms undergo assessment of their aerobic capacity and strength by the 6-minute walk test and handgrip dynamometry at baseline and at day 41. They also have a fasting blood draw and wear an actigraph for one week at baseline and week 6. Patients complete Functional Assessment of Chronic Illness Therapy-Fatigue and -Cognitive Subscales, Brief Fatigue Inventory, Multidimensional Fatigue Symptom Inventory, Center for Epidemiological Studies-Depression Scale State Trait Anxiety Inventory, Pittsburgh Sleep Quality Inventory, Profile of Mood States, Aerobic Center Longitudinal Study Physical Activity, and Symptom Inventory questionnaires at baseline and at day 41 and keep a daily exercise diary during study intervention.

ELIGIBILITY:
Inclusion criteria:

* primary diagnosis of cancer other than leukemia, with no distant metastasis
* chemotherapy naïve
* starting chemotherapy treatments for cancer and scheduled for at least 6 weeks of treatments with treatment cycles of either 2, 3 or 4 weeks. Oral chemotherapy (e.g., Xeloda) is acceptable
* Karnofsky Performance level of 70 or greater
* able to read English

Exclusion criteria:

* diagnosis of leukemia
* metastatic disease
* receiving concurrent radiation therapy
* physical limitations (e.g., cardiorespiratory, orthopedic, central nervous system) that contraindicate participation in a low to moderate intensity home-based walking and progressive resistance program
* identified as in the active or maintenance stage of exercise behavior as assessed by the Exercise Stages of Change Short Form

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 2009-09; Primary Completion 2016-02 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen M. Mustian, PhD, Principal Investigator — University of Rochester
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kleckner IR, Jusko TA, Culakova E, Chung K, Kleckner AS, Asare M, Inglis JE, Loh KP, Peppone LJ, Miller J, Melnik M, Kasbari S, Ossip D, Mustian KM. Longitudinal study of inflammatory, behavioral, clinical, and psychosocial risk factors for chemotherapy-induced peripheral neuropathy. Breast Cancer Res Treat. 2021 Sep;189(2):521-532. doi: 10.1007/s10549-021-06304-6. Epub 2021 Jun 30. PMID 34191201
- [Derived] Kleckner IR, Kamen C, Cole C, Fung C, Heckler CE, Guido JJ, Culakova E, Onitilo AA, Conlin A, Kuebler JP, Mohile S, Janelsins M, Mustian KM. Effects of exercise on inflammation in patients receiving chemotherapy: a nationwide NCORP randomized clinical trial. Support Care Cancer. 2019 Dec;27(12):4615-4625. doi: 10.1007/s00520-019-04772-7. Epub 2019 Apr 2. PMID 30937600
- [Derived] Kleckner IR, Kamen C, Gewandter JS, Mohile NA, Heckler CE, Culakova E, Fung C, Janelsins MC, Asare M, Lin PJ, Reddy PS, Giguere J, Berenberg J, Kesler SR, Mustian KM. Effects of exercise during chemotherapy on chemotherapy-induced peripheral neuropathy: a multicenter, randomized controlled trial. Support Care Cancer. 2018 Apr;26(4):1019-1028. doi: 10.1007/s00520-017-4013-0. Epub 2017 Dec 14. PMID 29243164
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/publications/pdq

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care + EXCAP | Standard Care
Started | 356 | 337
Completed | 331 | 312
Not Completed | 25 | 25
Not completed — Chemo started too soon | 2 | 3
Not completed — No Reason | 3 | 7
Not completed — Overwhelmed | 6 | 6
Not completed — Noncompliant | 1 | 4
Not completed — Medical | 1 | 3
Not completed — Changed Mind | 10 | 1
Not completed — Incomplete Form | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care + EXCAP | Standard Care | Total
Number analyzed (Participants) | 331 | 312 | 643
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (11.9) | 56.4 (10.1) | 56.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 306 | 298 | 604
  Male | 25 | 14 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity, Customized: White | 285 | 265 | 550
  Race/Ethnicity, Customized: Black | 30 | 30 | 60
  Race/Ethnicity, Customized: Other | 16 | 17 | 33
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg / m^2] — Measure Description: Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. Values below 18.5 represent "Underweight", 18.5 to 24.9 represent "Normal or Healthy Weight", 25.0 to 29.9 represent "Overweight" and 30.0 and above represent "Obese".
  kg / m^2 | 30.1 (6.7) | 30.2 (6.4) | 30.1 (6.5)
Currently Employed [Count of Participants; unit: Participants]
  Employed outside the house | 184 | 184 | 368
  Self-Employed | 11 | 16 | 27
  Home-Maker with >= 1 dependents | 32 | 23 | 55
  Unemployed | 104 | 89 | 193
Marital Status [Count of Participants; unit: Participants]
  Married or long-term committed relationship | 236 | 214 | 450
  Divorced or separated | 24 | 40 | 64
  Single | 44 | 36 | 80
  Widowed | 27 | 22 | 49
Education [Count of Participants; unit: Participants]
  Graduate degree | 67 | 46 | 113
  2 or 4 degree or Some college | 165 | 165 | 330
  High school / GED degree | 88 | 86 | 174
  No high school or GED degree | 10 | 14 | 24
  Unknown | 1 | 1 | 2
Cancer Type [Count of Participants; unit: Participants]
  Breast | 271 | 267 | 538
  Lymphoma | 17 | 7 | 24
  Colon | 20 | 15 | 35
  Lung | 6 | 9 | 15
  Other | 17 | 14 | 31
Cancer Stage [Count of Participants; unit: Participants] — Stage I.This stage is usually a small cancer or tumor that has not grown deeply into nearby tissues. It also has not spread to the lymph nodes or other parts of the body.
  Stage II and III.These stages indicate larger cancers or tumors that have grown more deeply into nearby tissue. They may have also spread to lymph nodes but not other parts of the body.
  Stage IV.This stage means that the cancer has spread to other organs or parts of the body. It may also be called metastatic cancer.
  Unknown Stage. There is not enough information to determine stage.
  Stage I is best, Stage IV is worst.
  Participants
    Stage I | 80 | 84 | 164
    Stage II | 150 | 139 | 289
    Stage III | 84 | 77 | 161
    Stage IV | 6 | 5 | 11
    Unknown | 11 | 7 | 18
Previous Treatment - Surgery [Count of Participants; unit: Participants]
  Yes | 296 | 275 | 571
  No | 35 | 37 | 72
Previous Treatment - Chemotherapy [Count of Participants; unit: Participants]
  Yes | 2 | 4 | 6
  No | 329 | 308 | 637
Previous Treatment - Radiation Therapy [Count of Participants; unit: Participants]
  Yes | 8 | 6 | 14
  No | 323 | 306 | 629
Previous Treatment - Hormone Therapy [Count of Participants; unit: Participants]
  Yes | 13 | 8 | 21
  No | 318 | 304 | 622
Time since end of first cancer treatment, weeks [Mean (Standard Deviation); unit: weeks] | 14.5 (72.9) | 6.8 (23.7) | 10.8 (55.2)
Karnofsky Performance Status (KPS) [Mean (Standard Deviation); unit: Karnofsky Performance Scale] — Measure Description: The Karnofsky Performance Scale (KPS) Index allows patients to be classified as to their functional impairment. Essentially as used in oncology, the KPS is a measure of time to death. A higher score is favorable. There are 3 general categories which are broken down into 11 specific criteria. Scale range is from 0 (Dead) to 100 (Normal, no complaints, no evidence of disease). The scale increases in units of 10.
  Karnofsky Performance Scale | 94.2 (7.1) | 94.8 (6.8) | 94.5 (7.0)
Exercise Stages of Change [Count of Participants; unit: Participants]
  Not exercising and don't intend to in next 6 month | 43 | 36 | 79
  Not exercising but do intend to in next 6 months | 89 | 83 | 172
  Not exercising but intend to in next 30 days | 199 | 192 | 391
  Exercising and have been for less than 6 months | 0 | 1 | 1
  Exercising and have been for more than 6 months | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change of Cancer-related Fatigue as Assessed by the Brief Fatigue Inventory (BFI) Total Score at Day 41 (After Exercise Intervention) Minus BFI Total Score at Day 0 (Before Exercise Intervention)
Description: BFI has nine items. Three items ask patients to rate the severity of their fatigue at its "worst," "usual," and "now" during normal waking hours, with 0 being "no fatigue" and 10 being "fatigue as bad as you can imagine." Six items assess the amount that fatigue has interfered with different aspects of the patient's life during the past 24 hours. The interference items include general activity, mood, walking ability, normal work (includes both work outside the home and housework), relations with other people, and enjoyment of life. The interference items are measured on a 0-10 scale, with 0 being "does not interfere" and 10 being "completely interferes." BFI Total Score is the average of the nine items, ranging from 0 (no fatigue) to 10 (high fatigue).
  The outcome measure is the change in the Brief Fatigue Inventory Total Score at day 41 (after exercise intervention) minus Brief Fatigue Inventory Total Score at day 0 (before exercise intervention).
Time Frame: 41 days: Day 0 (before intervention) Day 41 (post intervention)
Population: Subjects completing both BFI at day 0 and day 41
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care + EXCAP | Standard Care
Number analyzed (Participants) | 274 | 276
units on a scale | 0.9 (2.4) | 0.7 (2.3)
Statistical Analysis 1: Comparison: Standard Care + EXCAP vs Standard Care; Test type: Other; p = 0.9148, ANCOVA; Mean Difference (Final Values) = -0.01916, 95% CI 2-sided [-0.3710 to 0.3327], Standard Error of Mean 0.1791

ADVERSE EVENTS:
Arm/Group | Standard Care + EXCAP | Standard Care
Serious Adverse Events (participants affected / at risk) | 4/331 | 1/312
Other Adverse Events (participants affected / at risk) | 2/331 | 3/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Care + EXCAP (N=331) | Standard Care (N=312)
Lymphopenia, gr 4 leukocytes & neutrophils (Blood and lymphatic system disorders) | 1 | 0
Multi organ failure & susbsequent death (General disorders) | 1 | 0
Neutropenia & possible port infection (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia, cough, fever, fatigue (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Care + EXCAP (N=331) | Standard Care (N=312)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Failure to thrive (dehydra, hypokalemia, anorexia, diarrhea, fatigue (General disorders) | 1 | 0
Abdominal pain/acute typhilitis w/ neutropenia (Gastrointestinal disorders) | 0 | 1
Questionable thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0
Neutropenic fever (Blood and lymphatic system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No